CLINICAL TRIAL: NCT00601991
Title: A Multi-Center Phase 2 Study of Vascular Endothelial Growth Factor (VEGF) Trap as a Single Agent in Acute Myeloid Leukemia
Brief Title: A Multi-Center Phase 2 Study of VEGF Trap as a Single Agent in Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Another study was opened.
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephen Strickland, Assistant Professor of Medicine; Hematologist/Oncologist, Vanderbilt-Ingram Cancer Center
Masking: None | Purpose: Treatment
Other Study IDs: VICC HEM 0652; P30CA068485 (NIH); VU-VICC-HEM-0652; VU-VICC-061069
Record Dates: First submitted 2008-01-17; First posted 2008-01-28 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — aflibercept; Phlebotomy; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: VEGF Trap — Drug under investigation
  Other Names: Vascular endothelial growth factor trap
Procedure: Bone marrow biopsy — To determine response to treatment
Procedure: bone marrow aspiration — To determine response to treatment
  Other Names: Removal of a sample of bone marrow using a needle
Procedure: Venipuncture — For test of free VEGF Trap compared to bound VEGF Trap and for routine clinical testing during treatment
  Other Names: Taking blood sample

SUMMARY:
RATIONALE: Aflibercept may stop the growth of cancer cells by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying how well aflibercept works in treating patients with advanced refractory, relapsed, or untreated acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the response rate to aflibercept as a single agent in adult patients with advanced refractory, relapsed, or untreated acute myeloid leukemia (AML).
* To determine the 3-month progression-free survival following treatment with at least 4 courses of aflibercept in these patients.

Secondary

* To determine if there is any correlation between pre-treatment expression of VEGFR1 or VEGFR2 by marrow myeloblasts and disease response to aflibercept.
* To determine if bone marrow microvessel density (MVD) pre-treatment correlates with disease response to aflibercept, and if any decrease in MVD following treatment correlates with changes in bone marrow blast percentage (disease response).
* To assess changes in circulating endothelial cells (CEC) and circulating endothelial progenitor cells (EPC) as pharmacodynamic markers of aflibercept activity and possible correlates of disease response to aflibercept.
* To measure blood levels of free VEGF versus VEGF bound by aflibercept post-treatment to determine if the chosen dose of aflibercept is sufficient to bind all detectable soluble VEGF in these patients.
* To characterize the population pharmacokinetics of aflibercept with its associated interpatient variability and to explore for demographic and clinical covariates.
* To derive individual estimates of the duration over which VEGF-saturating aflibercept concentrations were systematically present and to examine their distribution across the population.
* To explore the potential relationship between the systemic-free and bound aflibercept levels and safety and efficacy data.

OUTLINE: This is a multicenter study.

Patients receive aflibercept IV over 1 hour on day 1. Treatment repeats every 14 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo bone marrow and blood sample collection periodically for pharmacokinetic/pharmacodynamic studies. Samples are analyzed for peak plasma-free aflibercept levels after the first infusion, trough plasma-free and bound aflibercept levels prior to each subsequent infusion and 60 days after the last infusion, and anti-aflibercept antibody via ELISA methods; circulating endothelial cells (CEC's) via ELISA and flow cytometry to determine if there is correlation between changes in circulating endothelial cells and changes in bone marrow blast percentage (i.e., disease response); myeloblast expression of VEGFR-1 and VRGFR-2 via immunohistochemistry (IHC); endothelial progenitor cells colony forming units (EPC-CFU's) to determine via in situ staining if changes in circulating endothelial progenitors following treatment with aflibercept correlates with disease response, and if there is a subpopulation of patients identified by pre-treatment circulating EPC-CFU's that may benefit from aflibercept; and bone marrow microvessel density (MVD) determination via immunohistochemistry.

After completion of study treatment, patients are followed for 60 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Acute myeloid leukemia (AML), as defined by WHO criteria and documented by morphologic examination of bone marrow aspirate and biopsy, including the following stages:

  * AML that is refractory to at least one course of induction chemotherapy
  * AML that has relapsed following one or more histologically documented complete remissions

    * Patients relapsing following chemotherapy alone, following autologous hematopoietic stem cell transplant, or following allogeneic hematopoietic stem cell transplant
  * Patients with untreated AML if they are felt not to be eligible for standard induction chemotherapy because of age or comorbidity
* No CNS disease

PATIENT CHARACTERISTICS:

Inclusion criteria:

* ECOG performance status 0-2
* Life expectancy ≥ 60 days
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 1.5 times ULN OR creatinine clearance ≥ 60 mL/min
* Urine protein:creatinine ratio < 1 OR 24-hour urine protein < 500 mg
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception prior to, during, and for at least 6 months after completion of study therapy

Exclusion criteria:

* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Serious or nonhealing wound, ulcer, or bone fracture
* History of allergic reactions attributed to compounds of similar chemical or biological composition to other agents used in the study
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of treatment
* Clinically significant cardiovascular disease within the past 6 months, including any of the following:

  * History of cerebrovascular accident
  * Myocardial infarction, coronary artery bypass graft, or unstable angina
  * New York Heart Association class III-IV congestive heart failure or serious cardiac arrhythmia requiring medication
  * Clinically significant peripheral vascular disease
  * Pulmonary embolism, deep venous thrombosis, or other thromboembolic event
* Uncontrolled hypertension, defined as BP > 150/100 mm Hg, or systolic BP > 180 mm Hg if diastolic blood pressure is < 90 mm Hg, on at least 2 repeated determinations on separate days within the past 3 months
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements
* Significant traumatic injury within 28 days prior to day 1 of therapy

PRIOR CONCURRENT THERAPY:

* Recovered from all therapy
* At least 4 weeks since prior chemotherapy and radiotherapy
* At least 4 weeks since prior FDA approved agents for treatment of myelodysplastic syndromes and/or AML, including lenalidomide and arsenic trioxide
* No prior anti-VEGF, anti-VEGFR, or antiangiogenic agents (e.g., bevacizumab)
* More than 28 days since prior major surgical procedure or open biopsy
* More than 2 days since prior bone marrow aspirate/biopsy or central venous catheter placement
* No anticipation of need for major surgical procedure during the study course
* Full-dose anticoagulation (e.g., warfarin) with PT/INR > 1.5 allowed provided that both of the following criteria are met:

  * In-range INR (usually between 2 and 3) on a stable dose of oral anticoagulant
  * No active bleeding or pathological condition that carries a high risk of bleeding (e.g., known varices)
* Prior and concurrent hydroxyurea allowed for blast control

  * Hydroxyurea must be discontinued no more than 24 hrs after the first dose of aflibercept
* No HIV-positive patients on combination antiretroviral therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03; Primary Completion 2009-03 (Estimated); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Response rate of aflibercept | day 14 of cycle 4 (14-day cycle)
  As determined by the International Working Group: Complete response: bone marrow blast(BMB) percentage (%) <=5% of nucleated cells and no detectable extramedullary disease; Partial response: BMB >5% but decreased by at least 50% pre-treatment (pre-tx) value OR extramedullary disease still present; Stable disease: BMB >5% and decreased or increased by <50% of pre-tx value and no new extramedullary disease; Progressive disease: BMB >=20% and an increase of at least 50% of pre-tx value and/or appearance of at least 50% in circulating blasts

SECONDARY OUTCOMES:
Bone marrow microvessel density determination at baseline, after courses 2 and 4 of treatment | at baseline, at day 29 and at day 57
  Density of microscopically small blood vessels in bone marrow biopsies
Pharmacokinetics of free versus bound VEGF Trap | Before and after 1st infusion on day 1, before infusion on day 1 of each 14-day cycle, and 60 days after last dose
  Blood levels of free VEGF Trap compared to bound VEGF trap to determine if the chosen level of VEGF Trap is sufficient to bind all detectable soluble VEGF in this group of patients
Progression-free survival in patients who achieve either a complete or partial response OR stable disease | at 12 weeks
  Patients who undergo a minimum of 4 cycles of treatment and who have either a complete or partial response to treatment or who have stable disease and who are free of progressive disease at 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Strickland, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center